CLINICAL TRIAL: NCT00545805
Title: Effects of the Surgical Removal of Visceral Fat Tissue (Omentectomy) on Insulin Sensitivity in Grade III Obese Volunteers Subjected to Bariatric Surgery
Brief Title: Surgical Removal of Visceral Fat Tissue (Omentectomy) Associated to Bariatric Surgery: Effects on Insulin Sensitivity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Marcelo Miranda de Oliveira Lima, MD, PhD, Marcelo Miranda de Oliveira Lima, MD, PhD, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIMED0001; FAPESP 05/58627-2
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Insulin Resistance; Obesity; Metabolic Syndrome X
Keywords: Insulin resistance; Metabolic syndrome X; Obesity; Intra-Abdominal Fat; Omentum; Bariatric surgery; Glucose Clamp Technique; Intravenous Glucose Tolerance Test; Adiponectin; Cytokines
MeSH Terms: conditions — Insulin Resistance; Obesity; Metabolic Syndrome | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OM group (Experimental)
  Interventions: Procedure: Roux-en-Y Gastric Bypass plus total omentectomy
- CT group (Active Comparator): Control group
  Interventions: Procedure: Roux-en-Y Gastric Bypass

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass plus total omentectomy — Roux-en-Y Gastric Bypass plus total omentectomy
  Arms: OM group
Procedure: Roux-en-Y Gastric Bypass — Roux-en-Y Gastric Bypass without omentectomy
  Arms: CT group

SUMMARY:
The intraabdominal fat is associated with insulin resistance, a condition that is in the basis of diabetes, metabolic syndrome and some cardiovascular diseases. It is not clear whether it is the origin of it or a surrogate marker only. We intend to compare the effects of bariatric surgery with versus without omentectomy in morbidly obese people intended to go through bariatric surgery, accessing insulin sensitivity by metabolic tests.

If the visceral fat is causative of insulin resistance, its surgical removal (omentectomy) might lead to improvement of insulin action, as seen in animal studies and in one study with morbidly obese human volunteers.

DETAILED DESCRIPTION:
In order to verify a potential additional benefit of omentectomy combined to Roux-en-Y silastic ring gastric bypass, insulin sensitivity will be studied by the gold-standard test, euglycemic-hyperinsulinemic clamp, since early postoperative follow-up (before significant weight variation), compared to a control group of bariatric surgery (same technique) alone. The variables will be analyzed in the post surgical evolution for correlation to metabolic changes: adiposity-related hormones and cytokines; lipid profile and other cardiovascular risk factors; molecular expression of biopsied subcutaneous adipocytes in vitro; anthropometrics; ultrasonography of abdominal subcutaneous and intra-abdominal fat depots and carotid intima-media thickness (preclinical atherosclerosis evaluation).

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 50 years.
* Female sex.
* BMI between 40 and 50kg/m2.
* Metabolic syndrome (NCEP/ATP III criteria).

Exclusion Criteria:

* Weight variation >5% within 3 months prior to preoperative tests.
* Use of antidiabetic medications within 3 months prior to preoperative tests.
* HbA1c >8%.
* Use of systemic corticosteroids for longer than 1 week within 3 months prior to preoperative tests.
* Hepatic cirrhosis, renal failure or any clinical condition (other than obesity) recognized as impairing insulin sensitivity.
* Present Smoking.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Increase of insulin sensitivity as measured by euglycemic-hyperinsulinemic clamp. | one month, six months and one year.

SECONDARY OUTCOMES:
increase of insulin secretion as measured by intravenous glucose tolerance test | one month, six months, one year
regression of carotid intima-media thickness | one month, six months, one year
Improvement of the insulin cell signalling in the subcutaneous adipose tissue. | one month, six months
increase of adipocytokines linked to greater insulin sensitivity and decrease of others linked to insulin resistance | one month, six months, one year

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo MO Lima, MD, Principal Investigator — University of Campinas (UNICAMP); Bruno Geloneze, PhD, Principal Investigator — University of Campinas (UNICAMP); José Carlos Pareja, PhD, Principal Investigator — University of Campinas (UNICAMP)
Locations (1):
- LIMED (Laboratory of Investigation of Metabolism and Diabetes)/GASTROCENTRO/Univeristy of Campinas (UNICAMP), Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Thorne A, Lonnqvist F, Apelman J, Hellers G, Arner P. A pilot study of long-term effects of a novel obesity treatment: omentectomy in connection with adjustable gastric banding. Int J Obes Relat Metab Disord. 2002 Feb;26(2):193-9. doi: 10.1038/sj.ijo.0801871. PMID 11850750
- [Background] Barzilai N, She L, Liu BQ, Vuguin P, Cohen P, Wang J, Rossetti L. Surgical removal of visceral fat reverses hepatic insulin resistance. Diabetes. 1999 Jan;48(1):94-8. doi: 10.2337/diabetes.48.1.94. PMID 9892227
- [Background] Gabriely I, Ma XH, Yang XM, Atzmon G, Rajala MW, Berg AH, Scherer P, Rossetti L, Barzilai N. Removal of visceral fat prevents insulin resistance and glucose intolerance of aging: an adipokine-mediated process? Diabetes. 2002 Oct;51(10):2951-8. doi: 10.2337/diabetes.51.10.2951. PMID 12351432
- [Background] Pitombo C, Araujo EP, De Souza CT, Pareja JC, Geloneze B, Velloso LA. Amelioration of diet-induced diabetes mellitus by removal of visceral fat. J Endocrinol. 2006 Dec;191(3):699-706. doi: 10.1677/joe.1.07069. PMID 17170226
- [Result] Lima MM, Pareja JC, Alegre SM, Geloneze SR, Kahn SE, Astiarraga BD, Chaim EA, Geloneze B. Acute effect of roux-en-y gastric bypass on whole-body insulin sensitivity: a study with the euglycemic-hyperinsulinemic clamp. J Clin Endocrinol Metab. 2010 Aug;95(8):3871-5. doi: 10.1210/jc.2010-0085. Epub 2010 May 19. PMID 20484482
- [Result] Lima MM, Pareja JC, Alegre SM, Geloneze SR, Kahn SE, Astiarraga BD, Chaim EA, Baracat J, Geloneze B. Visceral fat resection in humans: effect on insulin sensitivity, beta-cell function, adipokines, and inflammatory markers. Obesity (Silver Spring). 2013 Mar;21(3):E182-9. doi: 10.1002/oby.20030. PMID 23404948